CLINICAL TRIAL: NCT00003472
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Adult Patients With Oligodendroglioma
Brief Title: Antineoplaston Therapy in Treating Patients With Recurrent or Refractory Oligodendroglioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066509; BC-BT-17 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Oligodendroglioma, Adult
Keywords: Recurrent/progressive adult oligodendroglioma; Recurrent/progressive adult anaplastic oligodendroglioma
MeSH Terms: conditions — Oligodendroglioma; Recurrence | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Adults with a recurrent/progressive Oligodendroglioma will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for adult recurrent/progressive oligodendrogliomas provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of childhood brain tumors.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on adult recurrent/progressive oligodendrogliomas.

DETAILED DESCRIPTION:
OVERVIEW: This is a single arm, open-label study in which adults with recurrent/progressive oligodendrogliomas receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in adults with recurrent/progressive oligodendrogliomas, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in adults with recurrent/progressive oligodendrogliomas.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed incurable oligodendroglioma that progressed during or is recurrent or residual after initial therapy, including radiotherapy and/or chemotherapy
* Measurable tumor by MRI scan performed within two weeks prior to study entry
* Tumor must be at least 5 mm
* No brain stem tumors

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No severe heart disease
* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease (e.g., chronic obstructive pulmonary disease)

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections
* No other serious concurrent disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 4 weeks since prior immunotherapy

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* See Disease Characteristics
* At least 8 weeks since prior radiotherapy

Surgery:

* Recovered from any prior surgery

Other:

* No prior antineoplaston therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1996-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen patients were recruited between May 1996 and August 2007. All study subjects were seen at the Burzynski Clinic in Houston TX
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 13
Completed | 10
Not Completed | 3
Not completed — Not evaluable | 3

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: Years] | 41.5 [29.3 to 53.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 10
Participants
  Partial Response | 2
  Stable Disease | 4
  Progressive Disease | 4

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 13
Percentage of participants
  6 months overall survival | 76.9
  12 months overall survival | 61.5
  24 months overall survival | 46.2
  36 months overall survival | 23.1
  48 months overall survival | 15.4
  60 months overall survival | 7.7

ADVERSE EVENTS:
Time Frame: 11 years, 4 months
Description: Thirteen patients were recruited between May 1996 and September 2007. All study subjects were seen at the Burzynski Clinic in Houston TX
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 7/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=13)
Central Venous Catheter: Infection (General disorders) | 2 — The Central Venous Catheter: Infection were not related to Antineoplaston Therapy.
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 — The Fatigue (asthenia, lethargy, malaise) was not related to Antineoplaston Therapy.
Hemorrhage, CNS (Nervous system disorders) | 1 — The Hemorrhage, CNS was not related to Antineoplaston Therapy.
Infection (documented clinically): Blood (Infections and infestations) | 1 — The Infection (documented clinically): Blood was not related to Antineoplaston Therapy
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 1 — The Infection (documented clinically): Lung (pneumonia) was not related to Antineoplaston Therapy
Infection (documented clinically): Scrotum (Infections and infestations) | 1 — The Infection (documented clinically): Scrotum was not related to Antineoplaston Therapy.
Infection (documented clinically): Soft tissue NOS (Infections and infestations) | 1 — The Infection (documented clinically): Soft tissue NOS was not related to Antineoplaston Therapy.
Hypernatremia (Investigations) | 1 — The Hypernatremia was related to Antineoplaston Therapy.
Fracture (Musculoskeletal and connective tissue disorders) | 1 — The Fracture was not related to Antineoplaston Therapy.
Cognitive disturbance (Nervous system disorders) | 1 — The Cognitive disturbance was not related to Antineoplaston Therapy
Confusion (Nervous system disorders) | 1 — The confusion was related to Antineoplaston Therapy.
Neuropathy: motor (Nervous system disorders) | 1 — The Neuropathy: motor was not related to Antineoplaston Therapy
Seizure (Nervous system disorders) | 2 — The Seizures were not related to Antineoplaston Therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 — The Somnolence/depressed level of consciousness was not related to Antineoplaston Therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=13)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 4
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 4
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 2
Hypertension (Cardiac disorders) | 1
Central Venous Catheter: Infection (General disorders) | 4
Central Venous Catheter: Non-functional (General disorders) | 3
Central Venous Catheter: Pain (General disorders) | 1
Central Venous Catheter: Thrombosis/embolism (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 10
Fever (General disorders) | 1
Weight gain (General disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Edema/Fluid retention (General disorders) | 6
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam): Oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Hemorrhage, CNS (Nervous system disorders) | 1
Hemorrhage, GU: Bladder (Renal and urinary disorders) | 1
Infection - Other (Infections and infestations) | 1
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 2
Infection (documented clinically): Blood (Infections and infestations) | 1
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 2
Infection (documented clinically): Middle ear (otitis) (Infections and infestations) | 1
Infection (documented clinically): Mucosa (Infections and infestations) | 2
Infection (documented clinically): Scrotum (Infections and infestations) | 1
Infection (documented clinically): Soft tissue NOS (Infections and infestations) | 2
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 4
Infection (documented clinically): Urinary tract NOS (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 1
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1
Alkaline phosphatase (Investigations) | 2
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 2
Hypercholesteremia (Investigations) | 3
Hyperglycemia (Investigations) | 3
Hypernatremia (Investigations) | 6
Hypocalcemia (Investigations) | 4
Hypoglycemia (Investigations) | 3
Hypokalemia (Investigations) | 11
Hypophosphatemia (Investigations) | 3
Proteinuria (Investigations) | 2
SGOT (Investigations) | 1
SGPT (Investigations) | 1
Uric acid, serum-high (hyperuricemia) (Investigations) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 5
Mood alteration: Agitation (Nervous system disorders) | 1
Neurology - Other (Nervous system disorders) | 1
Pyramidal tract dysfunction (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 4
Somnolence/depressed level of consciousness (Nervous system disorders) | 6
Speech impairment (Nervous system disorders) | 3
Neuropathy: motor (Nervous system disorders) | 1
Ocular/Visual - Other (Eye disorders) | 1
Pain: Abdomen NOS (Gastrointestinal disorders) | 1
Pain: Bladder (Renal and urinary disorders) | 1
Pain: Breast (Endocrine disorders) | 1
Pain: Chest wall (Musculoskeletal and connective tissue disorders) | 1
Pain: Head/headache (Nervous system disorders) | 8
Pain: Joint (Musculoskeletal and connective tissue disorders) | 1
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 3
Pain: Neck (Musculoskeletal and connective tissue disorders) | 1
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No